CLINICAL TRIAL: NCT07187011
Title: Phase 2a Trial: Efficacy and Safety of PT150 in the Treatment of US Veterans With Posttraumatic Stress Disorder (PTSD)
Brief Title: Initial Study Sesting Efficacy and Tolerability of PT150 for PTSD in Veterans
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: San Diego Veterans Healthcare System (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); Pop Test Oncology LLC (Industry)
Responsible Party: Principal Investigator, Victoria Risbrough, VA Research Career Scientist/Health Science Research Specialist/Professor of Psychiatry, San Diego Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H250195; HT94252510832 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: glucocorticoid; cortisol; trauma; veteran; PT150
MeSH Terms: conditions — Combat Disorders; Wounds and Injuries | interventions — (11R,13S,17S)-11-(1,3-benzodioxol-5-yl)-17-hydroxy-13-methyl-17-prop-1-ynyl-1,2,6,7,8,11,12,14,15,16-decahydrocyclopenta(a)phenanthren-3-one

STUDY DESIGN:
Intervention Model Description: Intervention model: The investigators propose a two-site parallel group, randomized, double-blind, placebo-controlled Phase IIa clinical trial to test the efficacy and safety of PT 150-900 mg daily for 14 days for PTSD symptoms in Veterans.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- PT150 (Experimental): 150-900 mg study drug dose titrated over 7 days
  Interventions: Drug: PT150

INTERVENTIONS:
Drug: PT150 — Glucorticoid antagonist 900 mg
  Arms: PT150
Drug: Placebo — 900 mg
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the drug PT150, which blocks glucocorticoid receptor (GR) signaling, for treatment of PTSD in Veterans, and establish a safety and efficacy profile that will inform the design of future studies.

DETAILED DESCRIPTION:
This is a dual-site, proof-of-concept, parallel arm, double-blind placebo control study of a 14-day single daily dose of PT150/placebo in 100 Veterans with PTSD. Each site will enroll 60 Veterans with PTSD to ensure 100 study completers. Preclinical studies of PT150 and similar types of glucocorticoid antagonists have shown that they block stress responses in both acute and chronic models of stress response. PT150 has been tested previously in healthy control populations and in populations with depression, with it being found to be well tolerated and safe. Drug interaction results suggest it does not interact with alcohol or serotonin reuptake inhibitors, again supporting its safety and making it a candidate for further development. The goal of this Phase2a study is to tests its efficacy to reduce PTSD symptoms, as well as other biomarkers associated with PTSD. Participants first will undergo screening procedures, including a medical exam, clinical interview, self-report questionnaires, and blood draw. If eligible, they will be randomized to either PT150 or placebo. The PT150 dose will be titrated from 150-600mg over days 1-7, with the max dose of 900mg/day given the remaining 7 day timeframe. The same procedures will be repeated before, during and after taking the study drug or placebo for fourteen days. The key outcome measures will be obtained at baseline, day 28, and day 84.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Be a military service member or Veteran
* Male or female, 18-65 years of age
* Meet DSM-5 criteria for PTSD ≥ 3 months duration as determined by CAPS-5
* Normal vitals and a baseline EKG with clinically normal sinus rhythm, clinically normal conduction, normal QTc, and no clinically significant arrhythmias
* Self-reported medical history and brief physical examination with no clinically significant contraindications for study participation
* Blood laboratory test results for routine hematology, chemistries, liver and kidney function tests within acceptable limits
* Willing to comply with all study procedures including taking oral medication, the study schedule and be available for the duration of the study Biological females, if able to conceive, must agree to use 2 forms of non-hormonal, medically acceptable contraception.

Exclusion Criteria:

* Severe alcohol or substance use disorders by DSM-5 criteria in past 3 months or positive urine test for substances other than cannabis
* History or diagnosis of neurodegenerative disorders, psychotic disorders or bipolar disorder. Current treatment with antipsychotic medication for mental health
* History of suicide attempts and/or current suicidal ideation with plan or intent
* Currently using psychotropic medication (except SSRI/SNRI) or other drugs or agents which might interact with study drug. Currently taking SSRI/SNRI antidepressants for less than 30 days. Benzodiazepines or sleep agents (e.g. eszopiclone; zolpidem) are excluded; exception: trazodone 25-50 mg qhs prn for sleep or prazosin for nightmares
* Be pregnant or nursing
* HRT dose not stable for a minimum of 3 months
* Evidence of a serious, chronic medical condition that would increase the risk of an adverse outcome or history of any serious metabolic or other disease known to affect the CNS
* Have evidence of untreated or unstable medical illness including cardiovascular, neuroendocrine, autoimmune, renal, hepatic, or active HIV+/AIDS infection
* Serious cognitive impairment likely to interfere with ability to meaningfully participate
* Past brain injury/head trauma with minor loss of consciousness and current symptoms or significant loss of consciousness
* Current signs of violence or aggression
* A history of adrenal insufficiency or a plasma cortisol level ≤ 5 mcg/dl at screening
* Receiving non-pharmacotherapy treatments or procedures for where precautions exist for taking with PT150 and/or those that might interfere with the study
* Contraindication(s) to take PT150 such as renal or hepatic impairment, congenital metabolic disorders, or hypersensitivity to study drug or similar compounds
* Participation in a pharmaceutical trial or use of investigational drugs within 1 month of screening
* Hearing loss that would interfere with the extinction recall measures
* Any other illness, condition, or use of medications which in the opinion of the PI and/or study investigator would preclude safe and/or successful completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptoms - Clinician Administered PTSD Scale for DSM-5 (CAPS) | approximately 4 weeks
  The CAPS is the gold standard assessment of PTSD, providing a dimensional and categorical measure of PTSD, and incorporates frequency and intensity of symptoms into a single severity score. This manualized clinician-assessed interview contains 30 items.

SECONDARY OUTCOMES:
Side Effects - Frequency, Intensity, Burden of Side Effects (FIBSER) | 1, 2, 4, 12 weeks post treatment initiation
  The FIBSER is a self-report 0-6 Likert-type scale that measures global frequency, intensity, and overall burden of side effects.
Alcohol Drinking - The Time Line Follow Back (TLFB) | 1, 2, 4 and 12 weeks after treatment initiation
  The Time Line Follow Back (TLFB) is designed for collecting self-reported, retrospective estimates of AOD use and is extensively used to assess daily AOD use in research and practice
PTSD Symptoms - follow up | 12 weeks post treatment initiation
  Clinician Administered PTSD Scale for DSM-5 (CAPS) will be administered at 12 weeks post treatment initiation to estimate longevity of effects of PT150 on PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Risbrough, PhD, Principal Investigator — San Diego VA Healthcare System
Locations (2):
- United States (2):
  - Jennifer Moreno Department of VA Medical Center, San Diego, California
  - Michael E DeBakey VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
We plan on sharing the de-identified data (self report, clinician assessments, laboratory measures) with qualified investigators through the National Institute of Mental Health Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be provided 1 year after study completion.
Access Criteria: NDA-approved research investigators will be able to access the data.